CLINICAL TRIAL: NCT04922346
Title: The Relationship Between Physical Activity Level and Fear of Birth (Tokophobia) in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ali Omer Acar, Physiotherapist, Marmara University
Other Study IDs: E-18457941-050.99-10607
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Fear of Childbirth
Keywords: pregnancy; fear of childbirth; tokophobia; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Pregnant: All volunteer pregnant women who were in the 2nd and 3rd trimesters (between 14-40 weeks) and who met the inclusion criteria in the study

SUMMARY:
The aim of this study is to determine the effects of physical activity on fear of childbirth (tokophobia) in pregnant women.

DETAILED DESCRIPTION:
Fear of childbirth is defined as the fear felt and experienced before, during and after birth. Fear of childbirth is an acceptable level of fear and motivates the woman to prepare for the birth. However, if the fear developed before pregnancy and/or the severity of the fear increased during pregnancy, this situation is called "Tokophobia".

Physical activity is defined as body movements that are performed by using the body's muscles and joints, require energy expenditure above the basal level, can be performed at different intensities, increase heart rate and respiration, and occur with the contraction of large muscle groups.

It has been shown in the literature that physical activity in pregnant women contributes to the health of both the mother and the infant.

Several studies have reported the benefits of physical activity and exercise in preventing many risks of pregnancy, including lowering the risks of excess weight gain, preeclampsia, gestational diabetes, gestational hypertension, prenatal depression and macrosomia, and improving psychological well-being.

Despite the reported benefits of regular physical activity in the literature, it has been reported that the level of physical activity during pregnancy is lower compared to the pre-pregnancy period.

ELIGIBILITY:
Inclusion Criteria:

Having difficulty in communicating in order to understand and answer the evaluation questions correctly, Being at 14-40 weeks of gestation, Pregnancies with regular perinatal control.

Exclusion Criteria:

Being chronically ill or obese Individuals with a history of orthopedic, neurological, rheumatological or cardiopulmonary disease or surgery, Having 2 or more miscarriages, Multiple pregnancy, High-risk pregnancy Continuous vaginal bleeding Pre-pregnancy Body Mass Index (BMI) less than 17.5.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Wijma Delivery Expectation/Experience Scale (W-DEQ) | Baseline
  The "Wijma Delivery Expectation/Experience Scale (W-DEQ)" was developed by Klaas and Barbro Wijma, using the clinical experiences of women regarding the fear of childbirth. The W-DEQ scale version A was developed to measure the experiences of pregnant women before childbirth. Responses are on a six-point Likert-type scale from 0 to 5. 0 means "totally" and 5 as "not at all". While the minimum score on this scale is 0, the maximum score is 165. Higher scores indicate that women have a higher fear of childbirth.
The Pregnancy Physical Activity Questionnaire | Baseline
  The pregnancy physical activity questionnaire was developed by Lisa Chasan-Taber et al. in 2004 to determine the physical activity levels of pregnant women only. This questionnaire determines the activity level of pregnant women based on the time they spend during 32 activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Maltepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No